CLINICAL TRIAL: NCT06128525
Title: PRAMA (Prostate Resection After Microwave Ablation) MRI/Ultrasound Fusion Guided Transperineal Targeted Microwave Ablation for Prostate Cancer
Brief Title: Prostate Resection After Microwave Ablation (PRAMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4P-23-1; NCI-2023-02517 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-23-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2023-09-08; First posted 2023-11-13 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (TMA, radical prostatectomy) (Experimental): Patients undergo MRI/US fusion guided transperineal targeted TMA and then undergo standard of care RP same day or at 30 days post-TMA on study. Patients may undergo planning mpMRI of prostate prior to TMA. Patients also undergo blood sample collection at screening and post RP.
  Interventions: Procedure: Biospecimen Collection; Device: Microwave Ablation; Device: Multiparametric Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Radical Prostatectomy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Device: Microwave Ablation — Undergo transperineal MRI/US fusion guided transperineal targeted microwave ablation
  Other Names: Ablation, Microwave
Device: Multiparametric Magnetic Resonance Imaging — Undergo planning mpMRI of prostate
  Other Names: MP-MRI; mpMRI; Multi-parametric MRI; Multiparametric MRI
Other: Questionnaire Administration — Ancillary studies
Procedure: Radical Prostatectomy — Undergo RP
  Other Names: Prostatovesiculectomy

SUMMARY:
This phase I trial tests the safety of magnetic resonance imaging (MRI)/ ultrasound (US) fusion guided transperineal targeted microwave ablation (TMA) before a radical prostatectomy (RP) and how well it works in treating patients with prostate cancer. Prostate cancer is the second most common cancer in men and most will never become aggressive. Despite this, most men choose to undergo treatment which may include surgery. Removing the prostate gland and sometimes the lymph nodes (radical prostatectomy) is an invasive treatment for prostate cancer that can have a significant negative on quality of life. TMA is a less invasive procedure that uses high temperatures given through the skin between the scrotum and the rectum (transperineal). Using focused high energy and heating tumor cells to several degrees above normal body temperature may kill them without affecting the surrounding tissue. Using multiparametric (mp)MRI/US to create a 3-dimensional picture of the tumor may help in planning and preventing damage to healthy tissue. Giving MRI/US fusion guided transperineal TMA prior to radical prostatectomy may kill tumor cells, and may improve the quality of life in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of transperineal targeted microwave ablation of an MRI-identified index prostate cancer in patients undergoing radical prostatectomy.

SECONDARY OBJECTIVES:

I. KOELIS Trinity ability to plan and guide treatment needles and ablations in the prostate index lesion.

II. Impact of treatments on functional outcomes and quality of life. III. Predictability of Medwaves Avecure microwave ablation charts. IV. Predictability of post microwave ablation mpMRI.

OUTLINE:

Patients undergo MRI/US fusion guided transperineal targeted TMA and then undergo standard of care RP same day or at 30 days post-TMA on study. Patients undergo planning mpMRI of prostate prior to TMA. Patients also undergo blood sample collection at screening and post RP.

ELIGIBILITY:
Inclusion Criteria:

* Adult men diagnosed with prostate cancer and undergoing prostatectomy as treatment of choice
* Index lesion visible on multiparametric MRI confirmed by targeted biopsies using KOELIS Trinity (registered trademark)
* Patient suitable for intravenous (IV) sedation or general anesthesia and TMA
* Free, informed, and written consent, dated and signed before the enrollment and before any exam required by the trial

Exclusion Criteria:

* Past medical history of prostate surgery
* Past medical history of radiotherapy or pelvic trauma
* Past treatment for prostate cancer (PCa) (radiation, ablation, androgen deprivation therapy [ADT], chemotherapy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre Luis Abreu, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study opened in November 2023 and closed in August 2025. 1 subject was enrolled in the medical clinic at the University of Southern California, but withdrew consent and never began treatment nor study procedures. There was no data collected for this patient.
Period: Overall Study
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Patient withdrew consent | 1

BASELINE CHARACTERISTICS:
Population: 1 subject was enrolled, but withdrew consent and never began treatment nor study procedures. There was no data collected for this patient.
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: The Area of the Transperineal Targeted Microwave Ablation (TMA) Induced Tissue Death Assessed by Triphenyltetrazolium Chloride (TTC) Staining
Description: The excised prostate will be sliced at 4 mm intervals. Each slice will be embedded, and a pathologist will examine the slides corresponding to each slice. The pathologist will be blinded to MR and ultrasound imaging results. TTC staining is performed to determine the dead tissue induced by the TMA.
Time Frame: At time of radical prostatectomy (RP) immediately after TMA
Population: as for baseline characteristics
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of Adverse Events
Description: All adverse events graded according to the Clavien Dindo Classification
Time Frame: Up to 30 days after RP
Population: as for baseline characteristics
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Targeted Microwave Ablation (TMA) Procedure
Description: Measured by the probe-in/probe-out time and the ablation time.
Time Frame: At completion of TMA
Population: as for baseline characteristics
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Microwave Ablations Needed to Ablate One Multiparametric Magnetic Resonance Imaging (mpMRI)-Visible Lesion
Description: Count of microwave ablations needed to ablate one mpMRI-visible lesion will be reported
Time Frame: At time of TMA
Population: as for baseline characteristics
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 0

5. Secondary Outcome: The Area of the Transperineal Targeted Microwave Ablation (TMA) Induced Tissue Death Assessed by Hematoxylin and Eosin (H&E) Staining.
Description: The excised prostate will be sliced at 4 mm intervals. Each slice will be embedded, and a pathologist will examine the slides corresponding to each slice. The pathologist will be blinded to MR and ultrasound imaging results. H&E staining is performed to determine the dead tissue induced by the TMA.
Time Frame: At time of RP, 30 days after TMA
Population: as for baseline characteristics
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Difference Between the Ablation Location in the Prostate as Seen in the KOELIS 3-dimensional Map and the Ablation Location Observed Histologically on the Prostatectomy Specimen
Description: The difference between the ablation location as seen in the KOELIS 3D reconstruction of the prostate ("3D Map") will be compared to the ablation location observed histologically on the prostatectomy specimen.
Time Frame: Up to 1 month
Population: as for baseline characteristics
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Urinary Functions Assessed by International Prostate Symptoms Score and Uroflowmetry
Description: Urinary functions will be measured using International Prostate Symptoms Score (IPSS) and uroflowmetry. The IPSS can be 0-35 (higher score means worse urinary function). Uroflowmetry evaluates the maximum flow rate, average flow rate, flow time, voided volume, and the waveform of the flow rate.
Time Frame: At baseline and each follow up visit, up to 30 days after RP
Population: as for baseline characteristics
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Erectile Functions Assessed by International Index of Erectile Function-5 Score
Description: Erectile functions will be measured using International Index of Erectile Function (IIEF)-5 score. IIEF-5 score can be 5-25 (higher score means better erectile function).
Time Frame: At baseline and each follow up visit, up to 30 days after RP
Population: as for baseline characteristics
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Quality of Life Assessed by Expanded Prostate Cancer Index Composite-26 Short Form
Description: Quality of life (QOL) will be measured using Expanded Prostate Cancer Index Composite (EPIC)-26 Short Form score. EPIC-26 includes 13 questionnaires assessing several aspects of QOL. The interpretation of whether a higher numerical value in response to a questionnaire indicates a favorable outcome.
Time Frame: At baseline and each follow up visit, up to 30 days after RP
Population: as for baseline characteristics
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 0

10. Secondary Outcome: Difference Between the Treatment Effect Dimensions Measured Histologically on the Prostatectomy Specimen Resected After TMA, Compared to the Predictive Ablation Charts Provided by the Manufacturer
Description: The comparison of the difference between the treatment effect dimensions measured histologically on the prostatectomy specimen resected after TMA and the predictive ablation charts provided by the manufacturer will be performed.
Time Frame: Day after the TMA procedure
Population: as for baseline characteristics
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 0

11. Secondary Outcome: Difference Between the Treatment Effect Dimensions Measured Histologically on the Prostatectomy Specimen Resected One Month After TMA, Compared to Post TMA Dimensions Measured on the Pre-RP mpMRI
Description: The comparison between the treatment effect dimensions measured histologically on the prostatectomy specimen resected one month after TMA, compared to post TMA dimensions measured on the pre-RP mpMRI will be performed.
Time Frame: At time of RP, 30 days after TMA
Population: as for baseline characteristics
Arm/Group | Treatment (TMA, Radical Prostatectomy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days after last dose of study drug, up to 1.5 years.
Description: 1 subject was enrolled, but withdrew consent and never began treatment nor study procedures. There was no data collected for this patient.
Arm/Group | Treatment (TMA, Radical Prostatectomy)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT06128525/Prot_SAP_000.pdf